CLINICAL TRIAL: NCT04119596
Title: Study of the Genome, Gut Metagenome and Diet of Patients With Incident Parkinson's Disease
Status: Terminated | Type: Observational
Why Stopped: Low recruitment power
Sponsor: Atlas Biomed (Industry)
Responsible Party: Sponsor
Other Study IDs: PSM
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease; Genetic Predisposition
Keywords: Gut Microbiota; Parkinson's disease; Genetics; Microbiome; FFQ; GPAQ; HADS; MOCA
MeSH Terms: conditions — Parkinson Disease; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnosed Parkinson's disease: Patients with incident Parkinson's disease
  Interventions: Diagnostic Test: 16S rRNA gene sequencing; Genetic: DNA-microarray genotyping
- Control: Volunteers without diagnosed Parkinson's disease not meeting the exclusion criteria
  Interventions: Diagnostic Test: 16S rRNA gene sequencing; Genetic: DNA-microarray genotyping

INTERVENTIONS:
Diagnostic Test: 16S rRNA gene sequencing — Taking a stool sample for gut microbiome DNA sequencing
Genetic: DNA-microarray genotyping — Taking a saliva sample for genotyping

SUMMARY:
A case-control study to identify microbiome and genetic differences between healthy subjects and patients with incident Parkinson's disease.

DETAILED DESCRIPTION:
Two groups of subjects - one including healthy individuals and the other - treatment-naive patients with incident Parkinson's disease - will fill in the food frequency questionnaire, SF-36 questionnaire, HADS questionnaire and the physical activity questionnaire. All subjects must have 0-3 points on Hoehn and Yahr scale and more than 22 points on MoCA scale. DNA microarray genotyping will be used to process the DNA samples of the participants. The data on the composition of the participants' gut microbiota will be obtained through 16S rRNA sequencing of their stool samples.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 45 years and over who have been diagnosed with Parkinson's disease
* Subject signed informed consent

Exclusion Criteria:

* Gastroenterological diseases such as ulcerative colitis, Crohn's disease, celiac disease, gallbladder diseases (calculous cholecystitis, cholangitis, etc.) that are not related to functional disorders, a liver diseases or pancreas in medical history
* Exacerbations of chronic gastroenterological diseases
* Mental illness
* Oncology diseases
* Mental disorders
* Rheumatoid arthritis or other autoimmune diseases
* Acute infectious diseases or exacerbation of any diseases
* Recent (<3 months) administration of proton pump inhibitors, antimicrobial therapy or surgical intervention
* Recent (<3 weeks) use of probiotics, antacids, nonsteroidal anti-inflammatory drugs, laxatives
* Recent (<14 days) administration of laxatives (excluding prucaloprid)
* Recent (< 3 months) surgical intervention
* Pregnancy, planning to be pregnant or breast feeding at any point during the study or study enrollment
* Current alcohol/drug abuse (more than 3 points for women and 4 for men according to AUDIT-C questionnaire and/or more than 7 points on the AUDIT questionnaire) or addiction therapy within 12 months prior to screening
* Planned relocation from the home region during the study
* Stroke in medical history
* Any surgical intervention in the central nervous system
* Morbid obesity, BMI> 35 kg / m2
* A medical history of carriage or disease associated with a history of human immunodeficiency viruses, hepatitis B, C or Treponema pallidum
* The patient's inability to understand the essence of the study and agree to participate in it. MoCA scores <22
* 4-5 stage of the disease according to the Hen and Yara scale
* Severe somatic pathologies or any factors that, in the opinion of the doctor, may prevent the patient from being included in the study
* A medical history of serious head injuries
* Rheumatoid arthritis
* Tuberculosis

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients with incident Parkinson's disease from Russia
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Gut microbiome composition of participants | Baseline
  Bacterial relative abundance obtained via sequencing the DNA extracted from the stool sample
Genotypes of participants | Baseline
  High-throughput SNP profiling obtained via DNA-microarray genotyping of the DNA extracted from the saliva sample
Hoehn, Yahr scale | Baseline
  The Hoehn and Yahr scale defining five basic stages of PD progression (0-5)

SECONDARY OUTCOMES:
Physical activity questionnaire | Baseline
  Physical Activity Questionnaire - information on physical activity comprising 16 questions grouped in four domains: activity at work (1), travel to and from places (2), recreational activities (3), sedentary behaviour (4).
Food frequency questionnaire | 12 months before baseline
  Food frequency questionnaire assesses usual intake and portion size of more than 130 foods and beverages and more than 25 dietary supplements for the last 12 months. Responses are evaluated and analyzed to assess a dietary pattern for each group of subjects.
Change in Stool consistency | Baseline
  The Bristol stool scale is a diagnostic medical metric designed to classify the form of human faeces into seven categories
Change in Stool frequency | Baseline
  Change in the number of stool per week
Change in Quality of Life: SF-36 questionnaire | Baseline
  According to SF-36 questionnaire The Medical Outcomes Short-Form 36-Item Health Survey (SF-36) It is a self-administered questionnaire comprising 36-items measuring eight dimensions of general HRQOL: physical functioning (10 items), role limitation due to physical health problems (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), role limitations due to emotional problems (3 items), and general mental health (5 items). In addition to scores for individual dimensions, two summary scores assessing physical and mental dimensions of health and well-being can also be calculated: Physical Component Summary (PCS) score and the Mental Component Summary (MCS) score, respectively
Psychological distress questionnaire | Baseline
  Hospital Anxiety and Depression Scale (HADS) The aim of this study is to measure patients anxiety and depression, using the HADS : Hospital Anxiety and Depression scale.
  Scores of the HADS scale can be defined as:
  By adding the points of the answers: 1, 3, 5, 7, 9, 11, 13: we obtain the "Total A" which corresponds to the measure of the anxiety, then:
  7 or less: absence of symptomatology; 8 to 10: doubtful symptomatology; 11 and above: certain symptomatology.
  By adding the points of the answers: 2, 4, 6, 8, 10, 12, 14: we obtain the "Total B" which corresponds to the measure of the depression, then:
  7 or less: absence of symptomatology; 8 to 10: doubtful symptomatology; 11 and above: certain symptomatology. The minimal score is 0 and the maximal total score is 42
MOCA scale questionnaire | Baseline
  The MoCA assesses several cognitive domains:
  The short-term memory recall task (5 points) involves two learning trials of five nouns and delayed recall after approximately five minutes.
  Visuospatial abilities are assessed using a clock-drawing task (3 points) and a three-dimensional cube copy (1 point).
  Multiple aspects of executive functions are assessed using an alternation task adapted from the trail-making B task (1 point), a phonemic fluency task (1 point), and a two-item verbal abstraction task (2 points).
  Attention, concentration, and working memory are evaluated using a sustained attention task (target detection using tapping; 1 point), a serial subtraction task (3 points), and digits forward and backward (1 point each).
  Language is assessed using a three-item confrontation naming task with low-familiarity animals (lion, camel, rhinoceros; 3 points), repetition of two syntactically complex sentences (2 points), and the aforementioned fluency task.

CONTACTS AND LOCATIONS:
Locations (1):
- Siberian State Medical University, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No